CLINICAL TRIAL: NCT04341012
Title: Development of a Breath Analysis Test for Disease Diagnosis and Prognosis
Brief Title: Breath Analysis Based Disease Biomarkers
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tushar Patel, Principal Investigator, Mayo Clinic
Other Study IDs: 19-001971
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2024-11

CONDITIONS: Liver Diseases; Liver Cancer; COVID19
MeSH Terms: conditions — Liver Diseases; Liver Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal: No known medical conditions
  Interventions: Diagnostic Test: Collection of breath sample
- Liver Cirrhosis: Clinically diagnosed with cirrhosis
  Interventions: Diagnostic Test: Collection of breath sample
- COVID-19 tested: Persons with known test results for COVID-19 RNA
  Interventions: Diagnostic Test: Collection of breath sample
- Other: Persons with other medical diagnosis, no known liver disease, negative for COVID-19
  Interventions: Diagnostic Test: Collection of breath sample

INTERVENTIONS:
Diagnostic Test: Collection of breath sample — Analysis of volatile organic compounds in breath

SUMMARY:
The purpose of the study is to develop a clinical test based on breath analysis that can be used for disease diagnosis or prognosis.

DETAILED DESCRIPTION:
The study will seek to collect and analyze breath samples from a broad range of patients to develop reference ranges and to refine the testing methods. Protocols for breath sample collection and algorithms for analysis will be developed. Samples will be collected from normal volunteers, persons with documented liver disease, organ transplant or with known COVID-19 test results.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who are undergoing evaluation and obtaining clinical care at Mayo Clinic in Florida will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tushar Patel, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thomas JN, Roopkumar J, Patel T. Machine learning analysis of volatolomic profiles in breath can identify non-invasive biomarkers of liver disease: A pilot study. PLoS One. 2021 Nov 30;16(11):e0260098. doi: 10.1371/journal.pone.0260098. eCollection 2021. PMID 34847181

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from a specialized liver clinic. There was a need to ensure that sample collection and analysis could be performed within a controlled environment that did not pose risk of exposure or transmission of COVID-19 virus. As this could not be assured at the time, participants were not enrolled for the COVID-19 and other arms.
Groups:
- Healthy Patients: Patients with no known liver disease or cirrhosis
- Cirrhosis Patients: Patients with cirrhosis of the liver
Period: Overall Study
Arm/Group | Healthy Patients | Cirrhosis Patients
Started | 11 | 35
Completed | 11 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: sequentially enrolled patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Patients | Cirrhosis Patients | Total
Number analyzed (Participants) | 11 | 35 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 32 | 43
  >=65 years | 0 | 3 | 3
Age, Continuous [Median (Full Range); unit: years] | 45 [24 to 60] | 61 [33 to 76] | 57 [24 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 17 | 23
  Male | 5 | 18 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11 | 35 | 46
Number of subjects enrolled [Number; unit: participants] | 11 | 35 | 46

OUTCOME MEASURES:

1. Primary Outcome: Breath Volatile Organic Compound Profiles
Description: Detection of profiles of volatile organic compounds present in exhaled breath. The values in the table represent the number of participants from whom a volatile organic compound profile was able to be detected.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Patients | Cirrhosis Patients
Number analyzed (Participants) | 11 | 35
Participants | 11 | 35

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Healthy Patients | Cirrhosis Patients
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/35
Other Adverse Events (participants affected / at risk) | 0/11 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT04341012/Prot_000.pdf